CLINICAL TRIAL: NCT06765551
Title: Artificial IntelligenCe Based UlTrasonographic Assessment of IntensiVe CAre UniT-acquired WEakness (ACTIVATE)
Brief Title: AI Based Muscular Ultrasound to Assess Intensive Care Unit-acquired Weakness
Acronym: ACTIVATE
Status: Recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: University of Rostock (Other)
Responsible Party: Principal Investigator, Johannes Ehler, Principal Investigator, Jena University Hospital
Other Study IDs: 2024-3434-BO
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Unit-acquired Weakness; Artifical Intelligence; Ultrasound
Keywords: weakness; neuromuscular; critical illness polyneuropathy; critical illness myopathy; neuromuscular impairment
MeSH Terms: conditions — Asthenia; Polyneuropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with ICUAW (ICUAW+): Critically ill patients with ICUAW.
  Interventions: Diagnostic Test: Neuromuscular Ultrasound
- Patients without ICUAW (ICUAW-): Critically ill patients without ICUAW.
  Interventions: Diagnostic Test: Neuromuscular Ultrasound
- Healthy controls without ICUAW (ICUAW-)
  Interventions: Diagnostic Test: Neuromuscular Ultrasound

INTERVENTIONS:
Diagnostic Test: Neuromuscular Ultrasound — Non-invasive ultrasound of peripheral muscles of the upper and lower extremities with additional artificiall intelligence processing of ultrasound images.

SUMMARY:
The aim of this observational case-control study is to investigate, whether artificial intelligence can detect ultrasound-derived imaging characteristics typical for intensive care unit-acquired weakness. The main questions it aims to answer are:

1. Is the evaluation of specific parameters of neuromuscular ultrasound using AI-based image analysis suitable for detecting and monitoring critically ill ICU patients with ICUAW?
2. Do the results of AI-based ultrasound image analysis correlate with:

(A) the severity of ICUAW (B) the visual grading of muscle echogenicity (C) the 30- and 90-day-outcome?

DETAILED DESCRIPTION:
Intensive Care Unit-Acquired Weakness (ICUAW) is one of the most common neuromuscular complications in patients treated in intensive care. With increasing disease severity and especially in analgosedated, ventilated and delirious patients with limited ability to cooperate during the clinical examination, the detection and follow-up of ICUAW is limited to impossible. The clinical diagnosis and severity assessment of ICUAW is usually carried out with the help of established diagnostic methods (e.g. clinical-neurological examination, Medical Research Council-Sum Score, electrophysiological examinations), which, however, cannot be carried out regularly if the patient does not cooperate, thus delaying the diagnosis of ICUAW and making follow-up more difficult. Neuromuscular ultrasound (NMUS), on the other hand, is an easy-to-use, non-invasive examination option that is largely independent of patient compliance and is increasingly being investigated in patients with ICUAW. It was shown that NMUS can detect ICUAW and is helpful in assessing the severity of muscular weakness. However, the standardized recording and follow-up by means of scoring procedures (e.g. the 4-stage Heckmatt Scala) is assessed as partially subjective by the examiner and each individual ultrasound image must be taken with the human eye, taking into account various image parameters. To overcome these diagnostic limitations, artificial intelligence (AI) could be a useful extension or even an alternative.

AI is already being used in a variety of ways in medical diagnostics (e.g. in the detection of tumors and organ assessment), and increasingly also in the analysis of ultrasound images. In this study, the investigators aim to use AI, specifically Convolutional Neural Networks (CNNs), to classify ultrasound images into different categories based on muscle weakness. The main benefit of using AI for such tasks lies in the automation it provides. Once an AI model has been trained on an initial set of images, it can quickly categorize new, unseen images, significantly reducing the time and human effort required for diagnosis. AI models can analyze large amounts of data quickly and consistently, which is especially beneficial in a clinical intensive care setting. By applying AI, this study aims to train the detection and classification of muscle weakness in patients treated in intensive care. However, one challenge with AI models is their "black box" nature, where the decision-making process is not transparent. To solve this problem, the investigators will use explainable AI techniques (XAI) such as Grad-CAM (Gradient-weighted Class Activation Mapping) to visualize the specific areas of the ultrasound images that the AI model focuses on in its analysis. This not only helps validate the AI decisions, but also provides insights into the morphological changes in the muscles that come with different degrees of weakness.

By integrating AI and XAI, the study team aims to not only automate the detection and categorization of muscle weakness, but also improve our understanding of the underlying morphological changes in muscles. This dual approach could lead to more accurate and reliable diagnostics and ultimately improve outcomes for patients in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Major elective surgery, e.g. cardiothoracic or abdominal surgery
* Expected ICU stay >1 day postoperatively
* Healthy, age-machted subjects without ICUAW (recruited from staff of the department of anesthesiology and intensive care medicine)

Exclusion Criteria:

* No informed consent
* Emergency surgery
* Previous participation in the same study
* Preexisting neuromuscular disease
* Preexisting central nervous system disease with residual neuromuscular impairment (e.g. cerebral haemorrhage, stroke, brain tumor)
* High-dose glucocorticoid therapy (>300 mg hydrocortisone or equivalent per day) before or during particiation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with critical illness fulfilling the inclusion criteria should be screened for the study on two surgical ICUs at the department of anesthesiology and intensive care medicine of Jena University Hospital, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of abnormalities of muscle echogenicity assesed by muscular ultrasound | Day 14
  Determination of the number of patients correctly classified as ICUAW (+) using AI-based ultrasound evaluation

SECONDARY OUTCOMES:
Incidence of ICUAW severity assessed by Heckmatt Scale | Day 14
Incidence of ICUAW severity assessed by Medical Research Council Sum Score | Day 14
Days on ventilation | Day 30
Days on vasopressors | Day 30
Number of days in Hospital | Day 30
Number of patients with survival | Day 30
Frailty assessed by FRAIL-Scale | Day 30
Global outcome assessed by Bathel Index | Day 30
Number of patients with survival | Day 90
Frailty assessed by FRAIL-Scale | Day 90
Global outcome assessed by Bathel Index | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: PD Dr. Johannes Ehler, M.D., Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Jena University Hospital
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No